CLINICAL TRIAL: NCT04224441
Title: Repurposing the Antipsychotic Drug Chlorpromazine as a Therapeutic Agent in the Combined Treatment of Newly Diagnosed Glioblastoma Multiforme
Brief Title: Repurposing Chlorpromazine in the Treatment of Glioblastoma
Acronym: RACTAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marco G Paggi, MD, PhD (Other)
Collaborators: Regina Elena Cancer Institute (Other); Carlo Besta Neurological Institute (Other); Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor-Investigator, Marco G Paggi, MD, PhD, Medical Doctor, Clinical Pharmacologist, Regina Elena Cancer Institute
Organization: Regina Elena Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001988-75
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Glioblastoma Multiforme; MGMT-Unmethylated Glioblastoma
Keywords: drug repurposing; antipsychotic drugs; glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Chlorpromazine; Temozolomide

STUDY DESIGN:
Intervention Model Description: Addition of chlorpromazine to the standard GBM treatment during the adjuvant phase of the therapeutic protocol in un-methylated GBM patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard protocol plus chlorpromazine (CPZ) (Experimental): Combination of chlorpromazine to the standard treatment with temozolomide in the sole adjuvant phase of the standard protocol.Chlorpromazine will be administered at a dose of 50 mg/day concomitantly with the adjuvant treatment with temozolomide (TMZ)
  Interventions: Drug: Chlorpromazine Pill

INTERVENTIONS:
Drug: Chlorpromazine Pill — The experimental treatment involves the combination of chlorpromazine to the standard treatment with temozolomide solely in the adjuvant phase (after radio-chemotherapy, temozolomide for 5 days every 28, at a dose of 150-200 mg/mq for 6 cycles) of the Stupp protocol. Chlorpromazine will be administered at a dose of 50 mg/day concomitantly with the adjuvant treatment with temozolomide
  Other Names: Temozolomide

SUMMARY:
This study evaluates the addition of chlorpromazine to the first-line therapeutic protocol, i.e. maximal well-tolerated surgical resection followed by radiotherapy plus concomitant and adjuvant chemotherapy with temozolomide, in newly diagnosed glioblastoma multiforme patients carrying a hypo-methylated O6-methylguanine-DNA-methyltransferase (MGMT) gene

DETAILED DESCRIPTION:
Chlorpromazine (CPZ, Largactil, Thorazine) is a potent antagonist of the dopamine receptor D2 (DRD2) and has been effectively and safely employed for over half a century in the treatment of psychiatric disorders. CPZ displays a series of remarkable bio-molecular effects in cancer cells, as inhibition of cell growth, nuclear aberrations, inhibition of the phosphoinositide 3-kinase/mammilian target of rapamycin (PI3K/mTOR) axis, induction of cytotoxic autophagy, inhibition of glutamate and DRD2 receptors.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically-confirmed supra-tentorial GBM (World Health Organization grade IV) patients. Whenever feasible, patients will undergo maximal surgical resection or debulking, although patients with inoperable glioblastomas are also eligible.
2. Progression-free patients after having undergone maximal safe debulking surgery when feasible or biopsy, and
3. Patients undergone completed standard concomitant chemo-radiotherapy with temozolomide
4. Patients with provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
5. Patients (both males and females) should employ adequate contraceptive measures which should be maintained during the whole duration of the trial
6. Additional eligibility criteria include: age between 18 and 70; Karnofsky Performance Status (KPS) score of 70 or higher; adequate kidney, liver, bone marrow, and cardiac function; total serum bilirubin level and liver- function values; isocitrate dehydrogenase 1/2 (IDH1/2) mutational status; MGMT methylation status assessment.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria apply:

1. Treatment with any of the following:

   * Any other chemotherapy, immunotherapy or anticancer agents within 4 weeks before enrollment in the study.
   * Any investigational agents or study drugs from a previous clinical study within 30 days before the first dose of study treatment.
   * MGMT methylated
2. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including: uncontrolled hypertension; active bleeding diatheses; active hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV infection. Screening for chronic conditions is not required; inadequate bone marrow reserve or organ function, as demonstrated by laboratory parameters.

4. Judgment by the investigator that the patient should not participate to the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

5. Contraindications to MRI and or magnetic resonance spectroscopy (MRS). 6. Patients not able to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of toxicity | 6 months
  Toxicity evaluation of the combined treatment. Subjects will be evaluated for symptoms and adverse effects according to the NCI-CTCAE version 5.0 grading tool
Progression-free survival (PFS) | 6 months
  Effect of of adding CPZ to the standard GBM therapy, when compared with the standard therapy alone

SECONDARY OUTCOMES:
Evaluation of tumor response | 6 months
  Effect of of adding CPZ to the standard glioblastoma multiforme (GBM) therapy, when compared with the standard therapy alone
Overall survival (OS) | 6 months
  Effect of of adding CPZ to the standard glioblastoma multiforme (GBM) therapy, when compared with the standard therapy alone

CONTACTS AND LOCATIONS:
Overall Officials: Marco G Paggi, MD, PhD, Principal Investigator — Regina Elena Cancer Institute
Locations (3):
- Italy (3):
  - Regina Elena Cancer Institute, Rome, Lazio
  - Carlo Besta Neurological Institute, Milan, Lombardy
  - Istituto Oncologico Veneto, Padua, Veneto

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data describing primary and secondary outcomes will be made available
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available after 6 months after study completion
Access Criteria: Upon request. A valid Uniform Resource Locator (URL) will be reported

REFERENCES:
- [Background] Cohen BM, Lipinski JF. In vivo potencies of antipsychotic drugs in blocking alpha 1 noradrenergic and dopamine D2 receptors: implications for drug mechanisms of action. Life Sci. 1986 Dec 29;39(26):2571-80. doi: 10.1016/0024-3205(86)90111-6. PMID 2879204
- [Background] Nordenberg J, Fenig E, Landau M, Weizman R, Weizman A. Effects of psychotropic drugs on cell proliferation and differentiation. Biochem Pharmacol. 1999 Oct 15;58(8):1229-36. doi: 10.1016/s0006-2952(99)00156-2. PMID 10487524
- [Background] Pinheiro T, Otrocka M, Seashore-Ludlow B, Rraklli V, Holmberg J, Forsberg-Nilsson K, Simon A, Kirkham M. A chemical screen identifies trifluoperazine as an inhibitor of glioblastoma growth. Biochem Biophys Res Commun. 2017 Dec 16;494(3-4):477-483. doi: 10.1016/j.bbrc.2017.10.106. Epub 2017 Oct 21. PMID 29066348
- [Background] Lee MS, Johansen L, Zhang Y, Wilson A, Keegan M, Avery W, Elliott P, Borisy AA, Keith CT. The novel combination of chlorpromazine and pentamidine exerts synergistic antiproliferative effects through dual mitotic action. Cancer Res. 2007 Dec 1;67(23):11359-67. doi: 10.1158/0008-5472.CAN-07-2235. PMID 18056463
- [Background] Shin SY, Lee KS, Choi YK, Lim HJ, Lee HG, Lim Y, Lee YH. The antipsychotic agent chlorpromazine induces autophagic cell death by inhibiting the Akt/mTOR pathway in human U-87MG glioma cells. Carcinogenesis. 2013 Sep;34(9):2080-9. doi: 10.1093/carcin/bgt169. Epub 2013 May 20. PMID 23689352
- [Background] Barygin OI, Nagaeva EI, Tikhonov DB, Belinskaya DA, Vanchakova NP, Shestakova NN. Inhibition of the NMDA and AMPA receptor channels by antidepressants and antipsychotics. Brain Res. 2017 Apr 1;1660:58-66. doi: 10.1016/j.brainres.2017.01.028. Epub 2017 Feb 3. PMID 28167075
- [Background] Venkatesh HS, Morishita W, Geraghty AC, Silverbush D, Gillespie SM, Arzt M, Tam LT, Espenel C, Ponnuswami A, Ni L, Woo PJ, Taylor KR, Agarwal A, Regev A, Brang D, Vogel H, Hervey-Jumper S, Bergles DE, Suva ML, Malenka RC, Monje M. Electrical and synaptic integration of glioma into neural circuits. Nature. 2019 Sep;573(7775):539-545. doi: 10.1038/s41586-019-1563-y. Epub 2019 Sep 18. PMID 31534222
- [Background] Venkataramani V, Tanev DI, Strahle C, Studier-Fischer A, Fankhauser L, Kessler T, Korber C, Kardorff M, Ratliff M, Xie R, Horstmann H, Messer M, Paik SP, Knabbe J, Sahm F, Kurz FT, Acikgoz AA, Herrmannsdorfer F, Agarwal A, Bergles DE, Chalmers A, Miletic H, Turcan S, Mawrin C, Hanggi D, Liu HK, Wick W, Winkler F, Kuner T. Glutamatergic synaptic input to glioma cells drives brain tumour progression. Nature. 2019 Sep;573(7775):532-538. doi: 10.1038/s41586-019-1564-x. Epub 2019 Sep 18. PMID 31534219
- [Background] Zeng Q, Michael IP, Zhang P, Saghafinia S, Knott G, Jiao W, McCabe BD, Galvan JA, Robinson HPC, Zlobec I, Ciriello G, Hanahan D. Synaptic proximity enables NMDAR signalling to promote brain metastasis. Nature. 2019 Sep;573(7775):526-531. doi: 10.1038/s41586-019-1576-6. Epub 2019 Sep 18. PMID 31534217
- [Background] Caragher SP, Shireman JM, Huang M, Miska J, Atashi F, Baisiwala S, Hong Park C, Saathoff MR, Warnke L, Xiao T, Lesniak MS, James CD, Meltzer H, Tryba AK, Ahmed AU. Activation of Dopamine Receptor 2 Prompts Transcriptomic and Metabolic Plasticity in Glioblastoma. J Neurosci. 2019 Mar 13;39(11):1982-1993. doi: 10.1523/JNEUROSCI.1589-18.2018. Epub 2019 Jan 16. PMID 30651332
- [Derived] Pace A, Lombardi G, Villani V, Benincasa D, Abbruzzese C, Cestonaro I, Corra M, Padovan M, Cerretti G, Caccese M, Silvani A, Gaviani P, Giannarelli D, Ciliberto G, Paggi MG. Efficacy and safety of chlorpromazine as an adjuvant therapy for glioblastoma in patients with unmethylated MGMT gene promoter: RACTAC, a phase II multicenter trial. Front Oncol. 2023 Dec 14;13:1320710. doi: 10.3389/fonc.2023.1320710. eCollection 2023. PMID 38162492
- [Derived] Matteoni S, Matarrese P, Ascione B, Buccarelli M, Ricci-Vitiani L, Pallini R, Villani V, Pace A, Paggi MG, Abbruzzese C. Anticancer Properties of the Antipsychotic Drug Chlorpromazine and Its Synergism With Temozolomide in Restraining Human Glioblastoma Proliferation In Vitro. Front Oncol. 2021 Feb 26;11:635472. doi: 10.3389/fonc.2021.635472. eCollection 2021. PMID 33718225